CLINICAL TRIAL: NCT06402539
Title: The Effect of a Program Based on the Family-Centered Empowerment Model on Total Knee Prosthesis Patients and Their Caregivers: Randomized Controlled Study
Brief Title: Program Based on the Family-Centered Empowerment Model on Total Knee Prosthesis Patients and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Yasemin Sara, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 584847
Record Dates: First submitted 2024-04-16; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Caregiver
Keywords: total knee arthroplasty; Family Centered Empowerment Model; caregivers; care burden; self-efficacy; coping with stress; caregiving competence
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- receiving family-centered care (Experimental): IIn this randomized controlled clinical study, family-centered empowerment program (FCEM) will be implemented as an intervention. A total of 8 times (6 times face-to-face in the hospital; 2 times by phone) for 5 weeks. The content of face-to-face sessions consists of family-centered assessment, structured information booklet and bedside care skills training. Patients will be given a patient care booklet as part of this intervention.
  The content of the booklet; TKA surgery, preoperative period, postoperative period postdischarge care (daily tasks, surgical site care, weight gain, diet, driving, exercises It will include information enriched with visual materials regarding prevention of complications at home.
  The other part of the booklet consists of encouraging caregivers to actively participate in managing their own health and to maintain health-promoting behaviors such as nutrition, exercise, stress management and emotional management.
  Interventions: Behavioral: family-centered empowerment program
- waiting care group (No Intervention): Patients and families in the control group will be cared for according to the routine of the clinic and no intervention will be made.This group will be given a booklet on what to do after the last follow-up measurement, that is, after the 1st month post-operative check-up.

INTERVENTIONS:
Behavioral: family-centered empowerment program — The intervention will be carried out face to face in the Orthopedics and Traumatology outpatient clinic, and some interviews will be held by phone. The first interview is on the day the patient will be approved in the anesthesia department, the second interview is when the patient is admitted to the ward, the third interview is after the surgery and the fourth interview is in the ward on the day of discharge, the fifth interview is by phone 1 week after discharge, the sixth interview is at the outpatient clinic when the patient comes for a check-up 2 weeks after discharge, and the seventh interview is at the time of discharge. The eighth interview will be held by phone in the 3rd week after discharge, and the eighth interview will be held in the outpatient clinic in the 4th week after discharge.
  Arms: receiving family-centered care

SUMMARY:
In this study, the family empowerment model program given to individuals who underwent Total Knee Prosthesis and their caregivers was examined on the individuals' physiological function level, self-efficacy, and post-discharge hospital readmission (during the follow-up period); It was aimed to determine the effect of caregivers on their care burden, caregiving competence, and ability to cope with stress. The population of the research will consist of patients who underwent FFP surgery at Selçuk University Hospital Orthopedics and Traumatology Clinic between December 2023 and June 2024 and people who were cared for by the same family member for at least one month. The sample of the study will consist of patients and their caregivers who meet the inclusion criteria for the study. The sample of the study will consist of a total of 62 patients and their caregivers who were admitted to the clinic on the dates mentioned above and meet the inclusion criteria for the study. Study data will begin in the outpatient clinic and will be collected during the follow-up period until the 5th week after the patient is discharged. A training booklet created according to the Family-Centered Empowerment Model and a total of 9 sessions containing training and counseling will be applied to the intervention group of the study. Patients and families in the control group will be cared for according to the routine of the clinic and no intervention will be made. The data obtained will be analyzed using the IBM SPSS 25 (Statistical Packages for the Social Sciences - Undergraduate, Selçuk University) package program. Ethical principles will be observed at every stage of the study.

DETAILED DESCRIPTION:
Family involvement in perioperative education is beneficial to improve postoperative recovery outcomes and caregivers' experiences of patients after Total Knee or Hip Arthroplasty. Since patients are dependent on family members to meet their care needs immediately after discharge from the hospital after prosthetics, these individuals need to be equipped with sufficient knowledge and practical skills through education. Family members who provide quality care during recovery can contribute to reducing TKA/THA-related postsurgical complications and hospital readmissions and associated medical costs (e.g., ∼$20,000 per revision surgery).

In 2004, the Institute for Family Centered Care (IPFCC) defined family-centered care as mutually beneficial partnerships between healthcare providers, patients, and families in healthcare planning, delivery, and evaluation. Family-centered care has taken its place in the literature as a care model recommended to meet the needs of not only the patient but also the family members. The Family Centered Empowerment Model (FCEM) helps plan, implement and evaluate healthcare services through mutual partnerships of patients and families. Family-centered empowerment provides opportunities for family caregivers to gain knowledge and skills so that they can best manage family life and ultimately improve the lifestyles and quality of life of all family members. FCEM emphasizes individual agency and the role of other family members in three dimensions: motivational, psychological (self-esteem and self-control), and problematic individual characteristics (knowledge, attitudes, and perceived threat). Family empowerment has three main characteristics, including the ability to review necessary educational resources, the ability to make decisions and problem-solve, and the ability to communicate to meet current needs. Nurses play an important role by actively listening through reflective interaction to improve patients' understanding of their situation, problem-solving abilities, and control of their lives. Therefore, FCEM components are included in the nursing process. FCEM includes four main steps: (1) threat perception, (2) self-efficacy, (3) self-esteem, and (4) evaluation. Therefore, to achieve the best outcome, FCEM is expected to simultaneously increase knowledge, skills, values, and self-confidence and self-control beliefs in patients and their families. Studies have shown that ongoing education and empowerment of primary caregivers can significantly reduce patient readmission and mortality.

The effects of FCEM have been studied in various diseases. It has been proven that AMGM administration can improve the lifestyles of patients with heart failure. The effects of FCEM on reducing the care burden of caregivers of children with epilepsy and reducing perceived threats in heart failure patients have also been confirmed. However, only one study was found regarding the impact of using this model on caregivers of TKA and their family members. The results of this research show that adopting FCEM increases patient motivation and self-care effectiveness, promotes recovery of knee function in the short term after surgery, and reduces the likelihood of complications. There are gaps in the literature regarding the general experience and educational needs of family members of patients with TKA. First, previous research on caregivers' experiences has mostly used quantitative research methods and focused on caregiver burden. Secondly, it is thought that caregivers should be included in the research process to better understand the impact of TKA surgery on the caregivers of these patients. To improve the caregiving experience and ensure quality patient care, training that directly targets the needs of family caregivers should be implemented. There is limited research on supports such as family caregiver training or empowerment program after TKA.

ELIGIBILITY:
Inclusion Criteria: For patients :

* Being at least literate,
* Being 18 years or older,
* Ability to understand and speak Turkish,
* Having primary unilateral total knee arthroplasty surgery for the first time

The inclusion criteria for caregivers will be as follows:

* Volunteering for research,
* Being a relative of the patient (spouse, daughter, son-in-law, grandchild, daughter-in-law, son, brother, friend, etc.),
* Care for the patient for at least one month
* Being at least literate,
* Being 18 years or older,
* Ability to understand and speak Turkish,
* Being a caregiver to a patient with Total knee arthroplasty for the first time

Exclusion Criteria: for Patients

* Hearing and vision problems
* Mini mental test score below 25 points (less than 10 points indicate serious disorder, 10-19 points indicate moderate dementia, 19-24 points indicate early stage dementia).
* Having a communication problem such as vision or hearing that prevents the patient from understanding the information given and expressing it correctly.
* Having a diagnosed psychiatric disease

Exclusion Criteria for Caregivers

* Hearing and vision problems
* Mini mental test score below 25 points (less than 10 points indicate serious disorder, 10-19 points indicate moderate dementia, 19-24 points indicate early stage dementia).
* Having a communication problem such as vision or hearing that prevents the patient from understanding the information given and expressing it correctly.
* Having a diagnosed psychiatric disease,
* Providing paid care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Physiological function levels | Pre-test at the anesthesia clinic within 10 days before the surgery date. Post test on the 3rd day after surgery The last follow-up test was performed at the 4th week after surgery.
  Barthel Index:This scale evaluates mobility status and stair climbing functions such as feeding, washing, self-care, dressing, defecation control, urinary control, going to the toilet, ability to move from bed to wheelchair, walking or being dependent on a wheelchair, and stair climbing on a scale of 5-15 points (depending on the question). It consists of a total of 10 items that rate patients (0-15 points in 5-point increments). In this scale, the score that can be received is between 0-100, the higher the score, the more independent the patient is from other people and can manage his own business (0-20 points are fully dependent, 21- 61 points highly dependent, 62-90 points moderately dependent, 91-99 points mildly dependent, 100 points completely independent)

SECONDARY OUTCOMES:
Patient self-efficacy | Pre-test at the anesthesia clinic within 10 days before the surgery date. Post test on the 3rd day after surgery The last follow-up test was performed at the 4th week after surgery.
  General Self-Efficacy Scale:The score for each question varies between 1-5. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16 and 17 in the scale are reverse scored. The total score of the scale can vary between 17-85; An increase in the score indicates that self-efficacy belief increases.
  The increase in self-efficacy indicates that self-efficacy belief is increasing.
Readmission to the hospital within 30 days after discharge | Pre-test at the anesthesia clinic within 10 days before the surgery date. Post test on the 3rd day after surgery The last follow-up test was performed at the 4th week after surgery.
  30-day rehospital admission form (prepared by researchers):It will be monitored by asking an open-ended question whether there is a health problem that requires readmission due to any complications for 30 days after the surgery.
Care burden of caregivers | Pre-test at the anesthesia clinic within 10 days before the surgery date. Post test on the 3rd day after surgery The last follow-up test was performed at the 4th week after surgery.
  Zarit Caregiving Burden Scale:The scale evaluates the problems and care burden experienced by individuals providing care to individuals in need of care.
  The scale contains a total of 22 items and is a Likert-type scale in which each item is scored between 0 and 4. A score between 0 and 88 can be obtained from the scale. As the score obtained from the scale increases, the care burden experienced by the caregiver increases.
Caregiving competence | Pre-test at the anesthesia clinic within 10 days before the surgery date. Post test on the 3rd day after surgery The last follow-up test was performed at the 4th week after surgery.
  Caregiving Competence Scale: The degree of self-efficacy of the caregiver regarding the care of his/her patient is measured. The Likert type scale is arranged as ''1''=Not at all sufficient, ''2''=Somewhat sufficient, ''3''=Adequate and ''4''=Very sufficient. The lowest score from the scale is 4 and the highest score is 16. As the score obtained from the scale increases, the competence for caregiving increases.
Coping Response Inventory Scale | Pre-test at the anesthesia clinic within 10 days before the surgery date. Post test on the 3rd day after surgery The last follow-up test was performed at the 4th week after surgery.
  Participants gave the items in the inventory "5" if they always agree, "4" if they mostly agree, "3" if they sometimes agree, "2" if they rarely agree, "1" if they never agree. As a result of this scoring, while the maximum score to be obtained from an item is 5, the minimum score I 1. If the average score obtained from the inventory approaches 5, it shows that individuals have a high level of coping with stress.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Kurşun Kural, PhD, Study Director — Alanya Keykubat University; Fatma Taş Arslan, Professor, Study Director — Selcuk University
Locations (1):
- Selçuk University Faculty of Medicine Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' data will not be shared and will be archived by researchers.

REFERENCES:
- [Background] Larkin H. Poor accounting stymies HMO solvency audits. Hospitals. 1988 Nov 20;62(22):50. No abstract available. PMID 3181916
- [Background] Fields B, Rodakowski J, Leighton C, Feiler C, Minnier T, James AE. Including and Training Family Caregivers of Older Adults in Hospital Care: Facilitators and Barriers. J Nurs Care Qual. 2020 Jan/Mar;35(1):88-94. doi: 10.1097/NCQ.0000000000000400. PMID 30889081
- [Background] Gutenbrunner C, Stievano A, Nugraha B, Stewart D, Catton H. Nursing - a core element of rehabilitation. Int Nurs Rev. 2022 Mar;69(1):13-19. doi: 10.1111/inr.12661. Epub 2021 Jan 28. PMID 33506550
- [Background] Huang TT, Sung CC, Wang WS, Wang BH. The effects of the empowerment education program in older adults with total hip replacement surgery. J Adv Nurs. 2017 Aug;73(8):1848-1861. doi: 10.1111/jan.13267. Epub 2017 Mar 6. PMID 28122161
- [Background] Longo UG, Matarese M, Arcangeli V, Alciati V, Candela V, Facchinetti G, Marchetti A, De Marinis MG, Denaro V. Family Caregiver Strain and Challenges When Caring for Orthopedic Patients: A Systematic Review. J Clin Med. 2020 May 16;9(5):1497. doi: 10.3390/jcm9051497. PMID 32429398
- [Background] Manohar A, Cheung K, Wu CL, Stierer TS. Burden incurred by patients and their caregivers after outpatient surgery: a prospective observational study. Clin Orthop Relat Res. 2014 May;472(5):1416-26. doi: 10.1007/s11999-013-3270-6. PMID 24005979
- [Background] McIsaac DI, Beaule PE, Bryson GL, Van Walraven C. The impact of frailty on outcomes and healthcare resource usage after total joint arthroplasty: a population-based cohort study. Bone Joint J. 2016 Jun;98-B(6):799-805. doi: 10.1302/0301-620X.98B6.37124. PMID 27235523
- [Background] Mora-Traverso M, Molina-Garcia P, Prieto-Moreno R, Borges-Cosic M, Cruz Guisado V, Del Pino Algarrada R, Moreno-Ramirez P, Gomez-Jurado G, Gomez Tarrias C, Hidalgo Isla M, Jimenez Andres P, Linares Gago M, Lirola-Liebanas A, Mesa-Ruiz A, Munoz-Garach A, Salazar-Gravan S, Estevez-Lopez F, Martin-Matillas M, Ariza-Vega P. An m-Health telerehabilitation and health education program on physical performance in patients with hip fracture and their family caregivers: Study protocol for the ActiveHip+ randomized controlled trial. Res Nurs Health. 2022 Jun;45(3):287-299. doi: 10.1002/nur.22218. Epub 2022 Feb 11. PMID 35148434
- [Background] Provencher V, Clemson L, Wales K, Cameron ID, Gitlin LN, Grenier A, Lannin NA. Supporting at-risk older adults transitioning from hospital to home: who benefits from an evidence-based patient-centered discharge planning intervention? Post-hoc analysis from a randomized trial. BMC Geriatr. 2020 Mar 2;20(1):84. doi: 10.1186/s12877-020-1494-3. PMID 32122311